CLINICAL TRIAL: NCT03645499
Title: An Open-Label Study to Assess the Efficacy and Potential for Adrenal Suppression Following Maximal Use Treatment With TA-102 Topical Formulations in Subjects With Plaque Psoriasis.
Brief Title: An Open-Label Study to Assess Safety
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSTO 1723
Record Dates: First submitted 2018-08-21; First posted 2018-08-24 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Topical TA-102 A (Experimental): A thin layer of the study medication will be applied smoothly and evenly to affected areas (excluding face, axilla and groin areas) once daily
  Interventions: Drug: Topical TA-102 A
- Topical TA-102 B (Experimental): A thin layer of the study medication will be applied smoothly and evenly to affected areas (excluding face, axilla and groin areas) once daily
  Interventions: Drug: Topical TA-102 B
- Topical TA-102 C (Experimental): A thin layer of the study medication will be applied smoothly and evenly to affected areas (excluding face, axilla and groin areas) once daily
  Interventions: Drug: Topical TA-102 C
- Topical TA-102 D (Experimental): A thin layer of the study medication will be applied smoothly and evenly to affected areas (excluding face, axilla and groin areas) once daily
  Interventions: Drug: Topical TA-102 D
- Topical TA-102 E (Experimental): A thin layer of the study medication will be applied smoothly and evenly to affected areas (excluding face, axilla and groin areas) once daily
  Interventions: Drug: Topical TA-102 E

INTERVENTIONS:
Drug: Topical TA-102 A — applied smoothly and evenly to affected areas (excluding face, axilla and groin areas) once daily for 12 weeks
  Arms: Topical TA-102 A
Drug: Topical TA-102 B — applied smoothly and evenly to affected areas (excluding face, axilla and groin areas) once daily for 12 weeks
  Arms: Topical TA-102 B
Drug: Topical TA-102 C — applied smoothly and evenly to affected areas (excluding face, axilla and groin areas) once daily for 12 weeks
  Arms: Topical TA-102 C
Drug: Topical TA-102 D — applied smoothly and evenly to affected areas (excluding face, axilla and groin areas) once daily for 12 weeks
  Arms: Topical TA-102 D
Drug: Topical TA-102 E — applied smoothly and evenly to affected areas (excluding face, axilla and groin areas) once daily for 12 weeks
  Arms: Topical TA-102 E

SUMMARY:
An Open-Label study to assess safety

DETAILED DESCRIPTION:
An Open-Label study to assess the efficacy and potential for adrenal suppression following maximal use treatment with TA-102 topical formulations in subjects with Plaque Psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or non-pregnant female aged ≥ 18 years with a clinical diagnosis of plaque psoriasis.
2. Definite clinical diagnosis of stable plaque psoriasis for at least 6 months.
3. Subjects must be in good health and free from any clinically significant disease, including but not limited to, conditions that may interfere with the evaluation of plaque psoriasis.

Exclusion Criteria:

1. Female Subjects who are pregnant, nursing or planning to become pregnant during study participation.
2. History of allergy or sensitivity to retinoid, corticosteroids and/or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the Subject or the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
number of participants with adrenal suppression | 84 Days
  number of participants with adrenal suppression developed during the treatment with the study drug

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Yantovskiy, Study Director — Taro Pharmaceuticals Inc
Locations (1):
- Catawba Research, LLC, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No